CLINICAL TRIAL: NCT07173426
Title: Bioimpedance Integration for Optimized Fluid Management in Decompensated Heart Failure
Acronym: BIO-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 347894
Record Dates: First submitted 2025-03-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Decompensated Heart Failure
Keywords: Bioimpedance Analysis; Decompensated Heart Failure; Fluid Assessment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients admitted with decompensated Heart Failure are randomly allocated into one of the 2 groups using an online number generator:
  BIA Guided group In the BIA-Guided Group, BIA is performed within 24 hours of admission using a portable device that measures body water distribution and provides as estimated dry weight. These results, available within 2 minutes, help clinicians adjust diuretic therapy alongside standard assessments to achieve optimal fluid balance (euvolaemia).
  Standard Care Group In the Standard Care Group, BIA is performed by research staff and results are blinded from the clinical team. Fluid management relies on usual clinical judgement and diagnostic tools.
  All participants will receive follow-up 2-4 weeks after discharge, including NTproBNP blood tests, and the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) to evaluate heart failure symptoms.
  The investigators will then compare the primary outcome at 90 days in both these groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BIA-guided group (Active Comparator): Bioimpedance Analysis (BIA) will be performed within 24 hours of admission using the portable Bioscan touch i8 device (Maltron International, Essex, UK). The clinical team managing the patient will conduct serial BIA measurements and record the estimated dry weight in the patient's medical record during admission. Diuretic therapy and other fluid management strategies will be adjusted based on the BIA estimated dry weight throughout the hospital episode, in addition to standard clinical assessments, including physical examination and conventional diagnostic tools (e.g., chest X-ray, echocardiography), to achieve euvolaemia.
  Interventions: Device: Bioimpedance analysis
- Standard Care Group (No Intervention): A member of the research team not involved in the patients care will conduct the BIA and will record the estimated dry weight in the research records at enrolment (BIA 1) and at discharge (BIA 2). These results would be blinded to clinicians managing the patient, who will aim to achieve euvolemia based on usual clinical judgement, discretion and conventional diagnostic tools.

INTERVENTIONS:
Device: Bioimpedance analysis — Bioimpedance analysis involves electrodes attached to the patient's limbs which measures the resistance in the body to an imperceptible high-frequency, low-amplitude alternating electrical current. BIA measurements will include total body water (TBW), intracellular water (ICW), extracellular water (ECW), and the derived parameter "dry weight". Results are available at the bedside within 2 minutes.
  Arms: BIA-guided group

SUMMARY:
The goal of this clinical trial is to test whether using Bioimpedance Analysis (BIA) can help manage fluid levels in patients with heart failure who are admitted to the hospital with worsening symptoms. The main questions it aims to answer are:

1. Does BIA-guided fluid management reduce the need for extra treatment (in the form of diuretics which helps remove excess fluid from the body) or re-hospitalization for heart failure within 90 days after discharge?

Researchers will compare a group receiving BIA-guided treatment to a standard care group to see if BIA provides better results in managing fluid levels.

Participants will be randomly assigned to one of two groups:

BIA-Guided Treatment Group: Have BIA measurements done within 24 hours of admission and throughout their hospital stay to guide diuretic treatment.

Standard Care Group: Have BIA measurements taken at admission and discharge, but the results will not be shared with the clinical team, who will manage fluid levels as usual.

All patients will attend a follow-up visit in 2-4 weeks after discharge where the patient will undergo standard health checks, blood tests, and a questionnaire about how heart failure affects their quality of life.

The investigators will then compare both groups for the primary outcome measure, which is the rates of rehospitalisation or need for additional decongestive treatment, within 90 days of discharge from hospital.

DETAILED DESCRIPTION:
SCIENTIFIC RATIONALE Heart failure (HF) is a global health challenge affecting over 64 million people, with rising prevalence. Managing HF effectively is crucial to improving outcomes, but assessing and managing fluid status remains a significant challenge. Fluid congestion is a common cause of symptoms and hospitalizations for acute decompensated heart failure (ADHF). National audits indicate many patients are discharged before achieving adequate decongestion, increasing the risk of readmission and worsening prognosis.

Traditional methods, such as physical exams and imaging, correlate poorly with congestion. Conditions like obesity (BMI >30) and kidney disease further reduce the accuracy of diagnostic tools, including echocardiography and biomarkers like NT-proBNP. Hospitalizations for decompensated HF are associated with worse prognosis, progressive cardiac dysfunction, and higher mortality, highlighting the need for improved in-hospital management and prevention of readmissions.

Bioimpedance Analysis (BIA) is a promising non-invasive tool that measures body composition and fluid distribution, providing insights into total, intra-, and extracellular water. BIA is inexpensive, portable, and reproducible, making it suitable for regular clinical use. Studies suggest BIA-guided therapy may improve fluid management and reduce NT-proBNP levels, potentially enhancing outcomes.

This study aims to evaluate BIA's effectiveness in guiding fluid management in hospitalized HF patients with worsening symptoms. By enabling precise fluid assessment, BIA could optimize diuretic therapy and improve patient outcomes.

PRIMARY RESEARCH OBJECTIVE The principal research objective is to determine if BIA guided management of heart failure inpatients, compared to usual standard of care, results in a reduction in heart failure events within 90 days post discharge.

A heart failure event is defined as an outpatient requirement to increase oral diuretics or hospitalization for intravenous diuretics, due to decompensated heart.

SECONDARY RESEARCH OBJECTIVE

The secondary objectives are to determine if BIA guided management of heart failure inpatients, compared to usual standard of care, results in:

1. A higher rate of Acute Kidney Injury (defined by serum creatinine increase by (defined >=1.5 and <2 fold increase from baseline at any time)
2. A longer hospital Length of Stay including within a virtual ward.
3. A reduction in NTproBNP at 2-4 weeks after discharge from hospital.
4. An improvement in Patient Reported Outcomes (KCCQ-12), 2-4 weeks after discharge from hospital.
5. A lower rate of heart failure related events within 3, 6 months and 12 months.
6. A lower rate of All-cause mortality at 12 months

STUDY DESIGN This study is a single-centre, single-blinded, randomized controlled trial designed to evaluate the effectiveness of bioimpedance analysis (BIA) in guiding fluid management in patients who are hospitalized with acute decompensated heart failure (ADHF). The study aims to compare the outcomes of BIA-guided therapy versus standard care in terms of fluid management and HF-related outcomes.

PATIENT COHORT Eligible participants would include patients hospitalized for the management of Acute Decompensated Heart failure (ADHF), at Basildon and Thurrock University Hospital. All patients would be enrolled in the outpatients heart failure disease management programme.

Consent Potential participants will be identified and screened by the direct clinical team. If patients fulfil the eligibility criteria they will be approached by a member of their clinical care team. The clinical team will briefly explain the study and provide the patient with an ethically approved patient information sheet. This document will outline the details of the study, including its purpose, what participation involves, and how the patient's information would be used. The potential participants would be offered at least 24 hours to review the information and will have the opportunity to ask questions and consider whether they are interested in participating. This approach ensures that potential participants are introduced to the study by trusted healthcare professionals with whom they already have a clinical relationship. If the patient expresses interest and agrees, the research team can follow up to obtain formal consent and enrol the patient in the study. The original consent form will be retained in the site file, a copy provided to the patient and a copy inserted into the patient medical notes.

Randomization Participants provide consent will be randomized sequentially, in a 1:1 ratio using an online random number generator with an upper limit of 255, to either the BIA-guided therapy group or the standard care group. Odd-numbered patients will be assigned to the BIA-guided group (Group 1), and even-numbered patients will be assigned to the standard care group (Group 2).

Interventions BIA-Guided Group Bioimpedance Analysis (BIA) will be performed within 24 hours of admission using the portable Bioscan touch i8 device (Maltron International, Essex, UK). BIA measurements will include total body water (TBW), intracellular water (ICW), extracellular water (ECW), and the derived parameter "dry weight". Results are available at the bedside within 2 minutes. A member of the research team not involved in the patient's care will conduct the BIA and record the estimated dry weight in the patient's medical record. Diuretic therapy and other fluid management strategies will be adjusted based on the BIA estimated dry weight, in addition to standard clinical assessments, including physical examination, patient symptoms, and conventional diagnostic tools (e.g., chest X-ray, echocardiography), to achieve euvolaemia. BIA will also be performed at discharge for comparison to baseline results.

Standard Care Group A member of the research team not involved in the patient's care will conduct the BIA and will record the estimated dry weight in the research records at 24 hours of admission and at discharge. These results would be blinded to clinicians managing the patient, who will aim to achieve euvolemia based on usual clinical judgement, discretion and conventional diagnostic tools.

FOLLOW-UP All patients will be followed up in line with NICE guidelines for these patients, at 2-4 weeks post discharge. This will be conducted based on standard clinical assessments along with usual blood tests, to include NTproBNP. Furthermore, patients will be administered a quality-of-life questionnaire; Kansas City Cardiomyopathy Questionnaire (KCCQ-12); which is validated to assess symptoms, physical and social limitations, and quality of life in patients with heart failure, with respect to the preceding 2 weeks. Any additional contact with patients will be in line with routine clinical requirements. Outcomes will be recorded at pre-specified secondary endpoints.

SAMPLE SIZE CALCULATION 30-180-day readmission for heart failure is reported between 10-25%. The investigators have determined that a sample size of 232 (116 for each group) provides a two-sided 95% confidence interval for the difference in the event proportions with a width that is equal to 0.2. This provides a reasonable estimate of clinical significance for this pilot study when the estimated event proportion for the control group is 20% and 10% for the intervention group. The sample size was increased to 255 (an added 10%) to allow for some loss of information due to early study discontinuation.

DATA MANAGEMENT The data would be collected in an anonymized fashion and would be collated along with baseline demographic data as part of each hospital episode. The data would be analysed after 220 consecutive hospitalized patients have been entered into the study and each patient has been followed up for a minimum of 12 months.

STATISTICAL ANALYSES Statistical analyses would be performed using commercial software. A statistical significance level of 0.05 will be used. Discrete variables would be expressed as n (%) and continuous variables as mean (SD) or median (interquartile range [IQR]). Comparisons between survivors and non-survivors will be done with the use of chi-square test and Fisher exact test for categoric variables and t test for continuous variables if normally distributed or Mann-Whitney test if not normally distributed. The Spearman rank correlation would used to perform correlation analyses. All hypothesis testing will be 2 tailed. Cumulative incidences will be analysed by the method of Kaplan-Meier and compared using the log-rank test. In addition, the relationship between several clinical variables would be tested in a multivariate Cox model to predict long- term mortality and this will be described with hazard ratios (HR) and 95% Confidence Intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients with hospitalised with a decompensated episode of Heart Failure regardless of Ejection Fraction
3. Able and willing to consent.

Exclusion Criteria:

1. Patients on a palliative care pathway and/or estimated life expectancy <3 months
2. Patients admitted to ITU/ on intensive care support.
3. Patients currently taking part in any trials investigating new heart failure drug or interventional treatment.
4. Patients requiring Renal Replacement Therapy.
5. Patients unable or unwilling to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Event within 90 days post discharge | 90 days post discharge
  This is defined as outpatient requirement to increase oral diuretics or hospitalization for intravenous diuretics due to decompensated heart failure.

SECONDARY OUTCOMES:
Evidence of Acute Kidney Injury | At any time from hospitalisation till follow-up in Outpatient clinic 2-4 weeks after discharge
  Acute Kidney Injury is defined by ≥1.5 and <2 fold increase from baseline at any time.
Hospital Length of stay | 30 days
  The duration of hospitalization for patients with decompensated heart failure in both study arms.
NT pro-BNP after discharge from hospital | 2-4 weeks after discharge from hospital
  NT prob BNP levels will be measured during patient's outpatient follow-up visits in the Heart Failure clinic post discharge.
Patient Reported outcomes after discharge from hospital | 2-4 weeks post discharge
  Patients will be asked to complete the Kansas city Cardiomyopathy questionnaire during their Outpatient follow-up in the Heart Failure clinic 2-4 post discharge. This is to assess the severity of heart failure symptoms and their quality of life.
All-cause Hospitalisation at 3months | 90 days
  All-cause hospitalisations for patients in both groups (BIA guided and standard care groups) will be noted at 3 months.
All-cause Hospitalisation at 6 months | 6 months
  All-cause hospitalisations for patients in both groups (BIA guided and standard care groups) will be noted at 6 months.
All-cause hospitalisation at 12 months | 12 months
  All-cause hospitalisations for patients in both groups (BIA guided and standard care groups) will be noted at 12 months.
All-cause mortality at 12 months | 12 months
  All-cause mortality for patients in both groups (BIA guided and standard care groups) will be noted at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Basildon University Hospital, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santarelli S, Russo V, Lalle I, De Berardinis B, Vetrone F, Magrini L, Di Stasio E, Piccoli A, Codognotto M, Mion MM, Castello LM, Avanzi GC, Di Somma S; GREAT network. Prognostic value of decreased peripheral congestion detected by Bioelectrical Impedance Vector Analysis (BIVA) in patients hospitalized for acute heart failure: BIVA prognostic value in acute heart failure. Eur Heart J Acute Cardiovasc Care. 2017 Jun;6(4):339-347. doi: 10.1177/2048872616641281. Epub 2016 Apr 12. PMID 27073131
- [Background] Mayne KJ, Shemilt R, Keane DF, Lees JS, Mark PB, Herrington WG. Bioimpedance Indices of Fluid Overload and Cardiorenal Outcomes in Heart Failure and Chronic Kidney Disease: a Systematic Review. J Card Fail. 2022 Nov;28(11):1628-1641. doi: 10.1016/j.cardfail.2022.08.005. Epub 2022 Aug 28. PMID 36038013
- [Background] Alves FD, Souza GC, Clausell N, Biolo A. Prognostic role of phase angle in hospitalized patients with acute decompensated heart failure. Clin Nutr. 2016 Dec;35(6):1530-1534. doi: 10.1016/j.clnu.2016.04.007. Epub 2016 Apr 13. PMID 27118274
- [Background] Colin-Ramirez E, Castillo-Martinez L, Orea-Tejeda A, Vazquez-Duran M, Rodriguez AE, Keirns-Davis C. Bioelectrical impedance phase angle as a prognostic marker in chronic heart failure. Nutrition. 2012 Sep;28(9):901-5. doi: 10.1016/j.nut.2011.11.033. Epub 2012 Mar 30. PMID 22465907
- [Background] Di Somma S, Lalle I, Magrini L, Russo V, Navarin S, Castello L, Avanzi GC, Di Stasio E, Maisel A. Additive diagnostic and prognostic value of bioelectrical impedance vector analysis (BIVA) to brain natriuretic peptide 'grey-zone' in patients with acute heart failure in the emergency department. Eur Heart J Acute Cardiovasc Care. 2014 Jun;3(2):167-75. doi: 10.1177/2048872614521756. Epub 2014 Jan 29. PMID 24477201
- [Background] Di Somma S, De Berardinis B, Bongiovanni C, Marino R, Ferri E, Alfei B. Use of BNP and bioimpedance to drive therapy in heart failure patients. Congest Heart Fail. 2010 Jul;16 Suppl 1:S56-61. doi: 10.1111/j.1751-7133.2010.00162.x. PMID 20653713
- [Background] Massari F, Scicchitano P, Iacoviello M, Passantino A, Guida P, Sanasi M, Piscopo A, Romito R, Valle R, Caldarola P, Ciccone MM. Multiparametric approach to congestion for predicting long-term survival in heart failure. J Cardiol. 2020 Jan;75(1):47-52. doi: 10.1016/j.jjcc.2019.05.017. Epub 2019 Jul 17. PMID 31326239
- [Background] da Silva AT, Hauschild DB, de Almeida Oliveira LD, de Fragas Hinnig P, Franco Moreno YM, Wazlawik E. Association of hyperhydration evaluated by bioelectrical impedance analysis and mortality in patients with different medical conditions: Systematic review and meta-analyses. Clin Nutr ESPEN. 2018 Dec;28:12-20. doi: 10.1016/j.clnesp.2018.08.022. Epub 2018 Sep 21. PMID 30390867
- [Background] Sakaguchi T, Hirata A, Kashiwase K, Higuchi Y, Ohtani T, Sakata Y, Yasumura Y. Relationship of Central Venous Pressure to Body Fluid Volume Status and Its Prognostic Implication in Patients With Acute Decompensated Heart Failure. J Card Fail. 2020 Jan;26(1):15-23. doi: 10.1016/j.cardfail.2018.06.001. Epub 2018 Jun 9. PMID 29890212
- [Background] Jaffrin MY, Morel H. Body fluid volumes measurements by impedance: A review of bioimpedance spectroscopy (BIS) and bioimpedance analysis (BIA) methods. Med Eng Phys. 2008 Dec;30(10):1257-69. doi: 10.1016/j.medengphy.2008.06.009. Epub 2008 Aug 3. PMID 18676172
- [Background] Sakaguchi T, Yasumura K, Nishida H, Inoue H, Furukawa T, Shinouchi K, Miura H, Miyazaki K, Hamano G, Koide M, Abe H, Date M, Hirooka K, Koretsune Y, Kusuoka H, Yasumura Y. Quantitative Assessment of Fluid Accumulation Using Bioelectrical Impedance Analysis in Patients With Acute Decompensated Heart Failure. Circ J. 2015;79(12):2616-22. doi: 10.1253/circj.CJ-15-0723. Epub 2015 Oct 16. PMID 26477274
- See also: NICE guidance for diagnosis and management of chronic heart failure. — https://www.nice.org.uk/guidance/ng106
- See also: National Heart Failure Audit (NHFA) by National Institute for Cardiovascular Outcomes Research — https://www.nicor.org.uk/national-cardiac-audit-programme/heart-failure-audit-nhfa